CLINICAL TRIAL: NCT01110239
Title: Remote Ischemic Preconditioning to Ameliorate Delayed Ischemic Neurological Deficit After Aneurismal Subarachnoid Hemorrhage
Brief Title: Preconditioning for Aneurismal Subarachnoid Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sebastian Koch, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080406
Record Dates: First submitted 2010-04-21; First posted 2010-04-26 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Subarachnoid Hemorrhage
Keywords: limb preconditioning; remote preconditioning; ischemic preconditioning
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Ischemic Preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- remote limb preconditioning (Experimental): Subjects with subarachnoid hemorrhage will undergo escalating times of limb ischemia to determine tolerability and safety. The leg will be made transiently ischemic with application of a blood pressure cuff for up to 3 cycles of 10 minutes.
  Interventions: Procedure: remote limb preconditioning

INTERVENTIONS:
Procedure: remote limb preconditioning — 3 cycles of up to 10 minutes leg ischemia
  Other Names: ischemic preconditioning

SUMMARY:
In remote preconditioning, ischemia in one organ protects distant organs from ischemic insults. e.g. brief induced limb ischemia protects the brain from an otherwise more severe stroke.

The objective of this study is to determine if remote ischemic preconditioning can be safely and effectively instituted in patients with subarachnoid hemorrhage, who are at high risk for developing disabling cerebral ischemia. The investigators will also preliminarily assess if there is evidence for neuroprotection. This will be a Phase 1b study.

Additional objectives are:

1. to determine if remote ischemic preconditioning can be safely and effectively instituted in patients with subarachnoid hemorrhage, who are at high risk for developing disabling cerebral ischemia.
2. analogously to a dose-escalation study the investigators propose to study the safety and tolerability of increasing durations of limb ischemia until a target time of 10 minutes of limb ischemia has been reached.

DETAILED DESCRIPTION:
The investigators propose to study patients with subarachnoid hemorrhage, who generally have a high risk of ischemic stroke in the 2 weeks following the initial bleed, and patients with clipped or coiled aneurysm. The investigators will apply a blood pressure cuff around leg and use it to interrupt the circulation for 5-10 minutes. The investigators will repeat this for a total of 3 times every 24 to 48 hours up to 14 days. The cuff will be inflated for 5-10 minutes and then deflated for 5 minutes. There will be 3 cycles of this. The cuff will be inflated to 200mmHg.

The investigators will first start with 5 minutes of cuff inflation to either the arm or leg. The investigators will determine if this is safe in at least 6 patients. The investigators will then increase the duration of cuff inflation to 7.5 minutes for another 6 patients. If no adverse events are noted the investigators will the proceed to study 10 minutes of inflation in another 6 patients. If no side effects are noted the investigators will then determine that this is well tolerated.

The study will be monitored by a Data Safety Monitoring Board who will make decisions about escalating the duration of cuff inflation. If 2 or more patients develop an adverse event that is related to the procedure the investigators will stop and no longer continue at that level of cuff inflation and the previous level of cuff inflation will be determined to be the safe and tolerated level.

The investigators will collect safety data on adverse events such as tolerability, local tissue trauma or deep vein thrombosis.

ELIGIBILITY:
Inclusion Criteria: aneurismal subarachnoid hemorrhage

Exclusion Criteria:

1. Hunt Hess Scale > 4
2. Inability to undergo limb preconditioning due to local wound or tissue breakdown, history of peripheral extremity vascular disease or patient discomfort.
3. Inability to obtain informed consent from the patient or a health care proxy.
4. Ankle-brachial index < 0.7
5. Inability to start limb preconditioning within 4 days of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects admitted to a large community based teaching hospital were recruited between November 2008 and July 2010.
Groups:
- Sham Preconditioning: Subjects with subarachnoid hemorrhage will undergo escalating times of limb ischemia to determine tolerability and safety. The leg will be made transiently ischemic with application of a blood pressure cuff for up to 3 cycles of 10 minutes. A sham preconditioning group was added with only minimal cuff inflation.
Period: Sham Preconditioning
Arm/Group | Sham Preconditioning | 5-min Ischemia | 7.5-min Ischemia | 10-min Ischemia
Started | 7 | 14 | 7 | 6
Completed | 7 | 14 | 6 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: 5 Min Ischemia
Arm/Group | Sham Preconditioning | 5-min Ischemia | 7.5-min Ischemia | 10-min Ischemia
Started | 0 | 14 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 14 | 0 | 0
Period: 7.5 Min Ischemia
Arm/Group | Sham Preconditioning | 5-min Ischemia | 7.5-min Ischemia | 10-min Ischemia
Started | 0 | 0 | 7 | 0
Completed | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: 10 Min Ischemia
Arm/Group | Sham Preconditioning | 5-min Ischemia | 7.5-min Ischemia | 10-min Ischemia
Started | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Preconditioning: Subjects with subarachnoid hemorrhage will undergo escalating times of limb ischemia to determine tolerability and safety. The leg will be made transiently ischemic with application of a blood pressure cuff for up to 3 cycles of 10 minutes.
- Total: Total of all reporting groups
Arm/Group | Sham Preconditioning | 5 Min Ischemia | 7.5 Min Ischemia | 10 Min Ischemia | Total
Number analyzed (Participants) | 7 | 14 | 7 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9) | 53 (14) | 47 (12) | 62 (10) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 4 | 3 | 22
  Male | 1 | 5 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Deep Vein Thrombosis for Safety Assessment.
Time Frame: 90 days
Measure: Number; unit: participants
Groups:
- Sham Preconditioning: leg preconditioning with increasing durations of ischemia divided into 4 groups: sham preconditioning 3 cycles of 5min blood pressure cuff application 3 times 5 min cycles 3 times 7.5 min cycles 3 times 10 min cycles
Arm/Group | Sham Preconditioning | 5 Min Ischemia | 7.5 Min Ischemia | 10 Min Ischemia
Number analyzed (Participants) | 7 | 14 | 6 | 6
participants | 0 | 3 | 0 | 0

2. Primary Outcome: Visual Analog Scale Score as a Measure of Tolerability
Description: The visual analogue scale is a pain scale from 0-10, with 10 being maximum pain and is frequently used in research studies assessing patient discomfort.
Time Frame: 90 days
Population: We escalated the ischemia times in cohorts of 6. Cohorts of 6 were prespecified at the beginning to the study. All analysis was intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham Preconditioning: Limb preconditioning intervention at increasing durations of ischemia: 5, 7.5 and 10 min.
Arm/Group | Sham Preconditioning | 5 Min Ischemia | 7.5 Min Ischemia | 10 Min Ischemia
Number analyzed (Participants) | 7 | 14 | 6 | 6
units on a scale | 0 (0) | 3.6 (3.4) | 1.8 (2.1) | 2.5 (2.9)

ADVERSE EVENTS:
Arm/Group | Sham Preconditioning | 5 Min Ischemia | 7.5 Min Ischemia | 10 Min Ischemia
Serious Adverse Events (participants affected / at risk) | 3/7 | 9/14 | 1/7 | 1/6
Other Adverse Events (participants affected / at risk) | 5/7 | 8/14 | 3/7 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Preconditioning (N=7) | 5 Min Ischemia (N=14) | 7.5 Min Ischemia (N=7) | 10 Min Ischemia (N=6)
Delayed cerebral ischemia (Nervous system disorders) | 2 | 4 | 1 (1) | 0 (0)
low hematocrit (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
death (General disorders) | 0 | 1 | 0 | 0
ventriculitis (Infections and infestations) | 0 | 0 | 0 | 1
deep vein thrombosis (Vascular disorders) | 0 | 3 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Preconditioning (N=7) | 5 Min Ischemia (N=14) | 7.5 Min Ischemia (N=7) | 10 Min Ischemia (N=6)
hyponatremia (Metabolism and nutrition disorders) | 4 | 3 | 0 | 0
pneumonia (Infections and infestations) | 0 | 3 | 1 | 1
low hematocrit (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 1
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes